CLINICAL TRIAL: NCT00322166
Title: A Randomised Controlled Trial of Sunlight and Calcium Supplementation to Reduce Vitamin D Deficiency and Falls in Older People in Residential Care
Brief Title: The FREEDOM Study: a Randomised Controlled Trial of Sunlight and Calcium in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Prof Philip Sambrook, University of Sydney
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 402639; 0512-240M
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Accidental Falls
Keywords: accidental falls; vitamin D; parathyroid hormone; osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Sunlight; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A, Sunlight (Active Comparator): Participants in this arm are required to sit in the sun most days of the week for 15 minutes
  Interventions: Other: Sunlight
- Group B, sunlight and calcium (Active Comparator): Participants in this group receive sunlight and a calcium supplement
  Interventions: Other: Sunlight and calcium
- Group C (No Intervention): Control group
  Interventions: Other: control

INTERVENTIONS:
Other: Sunlight — Subjects in the intervention groups will be asked to undergo exposure of approximately 15% of their body (ie the face, hands and arms) usually between 9.30am - 10am daily during the year, 5 days per week.
  Arms: Group A, Sunlight
Other: Sunlight and calcium — Subjects in the intervention groups will be asked to undergo exposure of approximately 15% of their body (ie the face, hands and arms) usually between 9.30am - 10am daily during the year, 5 days per week. In the calcium and sunlight arm, calcium supplements (Caltrate, 600mg elemental calcium, Whitehall) will be administered to the whole group via the Blister/ Webster packs.
  Arms: Group B, sunlight and calcium
Other: control — Subjects in the control group will be provided with a brochure about vitamin D deficiency and how to treat it. They will receive their usual routine care and nutrition.
  Arms: Group C

SUMMARY:
The proposed study will determine the effect of a public health strategy (ie. increased sun light exposure and increased calcium intake) to reduce falls in older people in residential care using a randomised trial. The primary hypothesis of the trial is that increased appropriate sun light exposure will reduce falls, improve 25 hydroxy vitamin D (25OHD) levels and lower parathyroid hormone (PTH) levels. Secondary hypotheses are that the intervention will reduce accelerated bone turnover, reduce fractures, improve motor function and improve mood.

DETAILED DESCRIPTION:
Specific Aims and Objectives

The proposed trial will determine the effect of a public health strategy (ie increased sun light exposure and increased calcium intake) to reduce falls and fractures in older people living in residential care in a randomised trial. The primary hypothesis of the trial is that increased appropriate sun light exposure will reduce falls, improve 25OHD levels and lower PTH levels. Secondary hypotheses are that the intervention will reduce accelerated bone turnover, reduce fractures, improve motor function and improve mood.

Study Design

A randomised, controlled, multi-centre trial will be conducted over 12 months. Cluster randomization will be performed in hostels (low care residential aged care facilities) that agree to participate.

Participants

Participants will be recruited primarily from residential aged care facilities in Northern Sydney that have participated in the FREE study (currently 32 hostels). Men and women will be invited to participate in the study. Written informed consent from the participant or their proxy will be obtained.

The following general inclusion criteria will apply to subjects invited to participate:

* Aged 70 years or more
* Ambulant
* Likely to survive for more than 12 months, as assessed by the Implicit Review Tool employed in the FREE study
* Not taking vitamin D or calcium supplements
* No history of skin cancer in last three years

Interventions

Subjects in the intervention groups will be asked to undergo exposure of approximately 15% of their body (ie the face, hands and arms) usually between 9.30am - 10am daily during the year, 5 days per week. During mid summer, these sessions will run between 8.30am - 9am. It is recognised that it may be practically difficult to achieve this exposure during the months of June - August and exposure during these winter months may be less effective, but it considered important the study should run continuously through the year for adherence purposes. Adherence will be enhanced via the appointment of 'Sunlight Assistants' in each intervention institution, who will be normally employed in that institution for other duties but reimbursed for 1.5 hours per day for their duties in the study. During winter, late autumn and early spring or inclement weather, time lost will be made up during afternoon exposure on subsequent days. In the calcium and sunlight arm, calcium supplements (Caltrate, 600mg elemental calcium, Whitehall) will be administered to the whole group at the end of the sunlight exposure session. The Sunlight Assistants will record compliance with tablets.

Subjects in the control group will be provided with a facts sheet about vitamin D deficiency and how to treat it. They will receive their usual routine care and nutrition. All participants will receive the medical care usually provided by other health professionals.

Outcomes

Baseline data will be collected by study research staff, who will implement the intervention in each hostel initially, in conjunction with the Sunlight Assistants. Baseline measures will include demographic details, medication use, history of falls and fractures. Skin phenotype will be graded semi-quantitatively at baseline. UV tags will be used to measure actual exposure of hostel sunlight groups and examine dose -response relationships.

The primary outcome of falls will be assessed after the last cluster recruited has reached 12 months follow-up. Serum 25OHD and PTH will measured every 6 months to allow time trend and dose response analyses. Falls will be recorded by regular monthly visits to hostels including review of incident reports and clinical record review, as in the FREE study. Serum 25OHD will be measured using a specific radio-immunoassay with 100% cross-reactivity for 25OHD2 and 25OHD3 (DiaSorin Inc, USA). This assay has a sensitivity of 4nmol/L with an intra-assay precision of 7.6% and an inter-assay precision of 9.0% and was employed in the FREE study. Serum levels of intact PTH will also be determined as at baseline as in the FREE study by a two-site chemiluminescent enzyme-linked immunometric assay on a DPC Immulite 1000 analyser. This assay procedure measures the intact PTH molecule. The sensitivity of this assay is 1pg/ml and cross reactivity to PTH fragments and related compounds is low. The assay has a typical intra-assay precision of 5.5% and inter-assay precision of 7.9%. Biochemistry relevant to calcium metabolism including serum calcium, phosphate, albumin and creatinine will also be measured at baseline by standard autoanalyser methodology. Bone turnover will be measured using intact serum aminoterminal propeptide of type I procollagen (PINP) as a marker of bone formation and serum carboxyterminal telopeptide of type I collagen (CTX) as a marker of bone resorption, as employed in FREE. PINP will be determined using an automated immunoassay (Elecsys 170,__ Roche Diagnostics). This assay has a sensitivity of approximately 5 ng /mL with an intra-assay precision of approximately 2.3 %. CTX will be determined using an automated immunoassay (Elecsys 170_ Roche Diagnostics) with an intra-assay precision of approximately 2.0%. These turnover markers will be measured at baseline and 12 months.

Other secondary outcomes will include motor function measures related to falls risk (static balance, sit to stand test) assessed at baseline and 12 months using the same methodology employed in the FREE study. Quadriceps strength and body sway will also be assessed in a sub-sample. Fractures will be determined by regular visits (monthly) to hostels and validated by x-ray reports as in the FREE study. The effects of the intervention on mood will be assessed using the Geriatric Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or more
* Ambulant
* Likely to survive for more than 12 months, as assessed by the Implicit Review Tool employed in the FREE study
* Not taking vitamin D or calcium supplements
* No history of skin cancer in last three years

Exclusion Criteria:

* History of skin cancer in last three years
* Taking vitamin D or calcium supplements
* Not ambulant

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Falls | 1 year

SECONDARY OUTCOMES:
Vit D | 1 year
Fractures | 1 year
Geriatric Depression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philip Sambrook, MD, Principal Investigator — University of Sydney
Locations (1):
- Royal North Shore Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Sambrook PN, Cameron ID, Chen JS, Cumming RG, Durvasula S, Herrmann M, Kok C, Lord SR, Macara M, March LM, Mason RS, Seibel MJ, Wilson N, Simpson JM. Does increased sunlight exposure work as a strategy to improve vitamin D status in the elderly: a cluster randomised controlled trial. Osteoporos Int. 2012 Feb;23(2):615-24. doi: 10.1007/s00198-011-1590-5. Epub 2011 Mar 3. PMID 21369788